CLINICAL TRIAL: NCT01454453
Title: Rationalisation of Antipsychotic Drug Use in Older People, Using [18F]-Fallypride PET
Brief Title: Optimisation of Antipsychotic Drug Use in Older People
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Failure to recruit people with very late onset schizophrenia like psychosis
Sponsor: Institute of Psychiatry, London (Other)
Responsible Party: Principal Investigator, Suzanne Reeves, Clinician Scientist, Institute of Psychiatry, London
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2167SR
Record Dates: First submitted 2011-10-12; First posted 2011-10-19 (Estimated); Last update posted 2017-04-19 (Actual); Status verified 2017-04

CONDITIONS: Alzheimer's Disease; Schizophrenia
Keywords: amisulpride; receptor occupancy; antipsychotic sensitivity
MeSH Terms: conditions — Alzheimer Disease; Schizophrenia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Patients - dose titration (Experimental): Amisulpride 50-200mg, 4-12 weeks, with brain imaging
  Interventions: Drug: Patients- dose titration

INTERVENTIONS:
Drug: Patients- dose titration — dose titration (patients) - 4-10 weeks

SUMMARY:
Drugs such as amisulpride, known as antipsychotic drugs, are used to treat troublesome and distressing symptoms in older people. Although these drugs can be beneficial, they are associated with side effects, particularly in patients with dementia and schizophrenia- like illness. There is an urgent clinical need to understand why this is the case, to guide treatment strategies.

This study aims to utilise brain imaging techniques that measure the action of antipsychotic drugs in the brain to explore the causes of this susceptibility in older people with dementia and schizophrenia-like illness, and translate these findings into direct patient benefit.

The aim of the study is to investigate and compare the relationship between the action of amisulpride at brain sites during the first 10 weeks of amisulpride treatment in two patient groups - Alzheimer's disease and schizophrenia-like illness. Imaging data will be combined with data on drug dosage, levels of drug in the bloodstream and clinical response (symptom reduction and motor side effects) during dose titration.Dose-response modelling will be carried out in both groups to establish the minimum clinically effective dose of amisulpride, optimum dose range and impact of variability and covariates on exposure-response relationships

ELIGIBILITY:
Inclusion Criteria

Treatment and Control (antipsychotic free) Group

Schizophrenia

* meet diagnostic criteria for schizophrenia-like illness
* aged between 60 and 95 years of age
* score <6 on the Geriatric depression scale

Alzheimer's

* meet diagnostic criteria for AD
* score <=4 on the Modified Hachinski Ischaemia Scale
* score < 8 on a modified version of the UPDRS
* aged between 60 and 95 years of age
* score <6 on the Geriatric depression scale

Exclusion Criteria

Treatment Group

Schizophrenia

* current or past history of addiction, traumatic brain injury or epilepsy
* prescribed any drug that interferes with brain dopamine in past 2 weeks (6 weeks if depot antipsychotic medication).
* medical conditions that might affect Ability to tolerate a brain scan
* unable to give informed consent

Alzheimer's

* current or past history of psychiatric illness, traumatic brain injury or epilepsy
* prescribed an antipsychotic or other oral drug that interferes with brain dopamine function within the past 2 weeks (6 weeks if depot antipsychotic medication).
* medical conditions that might affect a person's ability to tolerate a brain scan

Control (antipsychotic free) Group

Schizophrenia

* Prescribed psychotropic medication
* unable to give informed consent

Alzheimer's

• Prescribed psychotropic medication

Ages: 60 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2012-05; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
dose titration | 12 weeks
  receptor occupancy compared across 2 patient groups following dose-titration

OTHER OUTCOMES:
modelling of dose-response relationships | 12 weeks
  dose-response modelling

CONTACTS AND LOCATIONS:
Overall Officials: Suzanne J Reeves, MBChB, PhD, Principal Investigator — Institute of Psychiatry, London
Locations (1):
- Institute of Psychiatry, Kings College London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No